CLINICAL TRIAL: NCT03318029
Title: A Systems Biology Approach to the Interaction Between Vitamin D Supplementation and Sunlight Exposure in Brazilian Women Living in Opposite Latitudes (The D-SOL Study).
Brief Title: Vitamin D Supplementation and Sunlight Exposure in Brazilian Women Living in Opposite Latitudes (The D-SOL Study)
Acronym: D-SOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Universidade Federal de Goiás (Unknown)
Responsible Party: Principal Investigator, Marcela Moraes Mendes, PhD Research Fellow, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D-SOL
Record Dates: First submitted 2017-10-11; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Supplementation; Sunlight
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: Two controlled, randomized, double-blind clinical trials developed and undertaken (one in Brazil and the other in the UK) with an intervention period of 12 weeks. The women selected were randomly divided into two groups: Placebo Group and Supplemented Group, the latter will receive 600UI of vitamin D, in each country. Groups (arms): Placebo UK trial; Vitamin D UK trial; Placebo Brazuk trial; Vitamin D Brazil trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo UK trial (Placebo Comparator): Placebo and living in the UK
  Interventions: Dietary Supplement: Placebo
- Vitamin D UK trial (Active Comparator): Vitamin D supplementation and living in the UK
  Interventions: Dietary Supplement: Vitamin D supplementation
- Placebo Brazil Trial (Placebo Comparator): Placebo and living in the Brazil
  Interventions: Dietary Supplement: Placebo
- Vitamin D Brazil Trial (Active Comparator): Vitamin D supplementation and living in Brazil
  Interventions: Dietary Supplement: Vitamin D supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin D supplementation — Vitamin D supplementation of 600 IU daily for 12 weeks
  Arms: Vitamin D Brazil Trial; Vitamin D UK trial
Dietary Supplement: Placebo — rice flour with no vitamin D
  Arms: Placebo Brazil Trial; Placebo UK trial

SUMMARY:
There is a consensus that vitamin D deficiency is a public health issue because of its implications in several diseases including, osteopenia, osteomalacia, heart disease, diabetes (type I and II), inflammatory diseases, multiple sclerosis and rheumatoid arthritis. Studies in sunny countries have shown that vitamin D deficiency is a common phenomenon, despite the abundance of sunlight in these places, which shows the influence of diet, skin pigmentation, cultural habits and also genetic factors on the metabolism of this vitamin. Thus, the study hypothesis is that vitamin D supplementation is required to obtain the optimal serum concentration in Brazilian people living both in Brazil and in the United Kingdom and that this response is dependent on the initial levels, being influenced by sunlight exposure, skin pigmentation, diet and polymorphisms of the vitamin D receptor gene. Two controlled, randomized, double-blind clinical trials were held (one in the UK and the other in Brazil) over a period of 12 weeks, with female subjects, Brazilian, aged 20 to 59 years. The women selected were divided into two groups: Placebo Group and Supplemented Group, the latter received vitamin D 600 IU. After the analysis of the effect of vitamin D supplementation compared to placebo, the investigators propose to analyse genome-wide transcriptomic expression in order to associate specific signal transduction and metabolic pathways to respective vitamin D responses. and a genetic risk score based on polymorphisms will be constructed. The 'systems level' approach will enable us to identify differences in gene expression and whether this explains why some individuals are 'good' responders or 'poor' responders to vitamin D supplementation. This is the first study that will examine two population groups of the same ethnic group and sex, living in different countries, with identical design studies. Our results first will determine how important supplementation and exposure to sunlight are for the serum level of vitamin D by comparing directly, using the same methodology, people living in different latitudes, as well as the genetic influence on the response to supplementation. The data will also provide both countries key data about the need to reconsider new revisions to dietary recommendations for vitamin D in adults.

DETAILED DESCRIPTION:
During this study the subjects were asked to visit the Clinical Investigation Unit, FHMS, University of Surrey in the UK or the Research Clinic, Faculty of Nutrition, Federal University of Goiás in Brazil, on two occasions, at the beginning of the study for baseline measurements and at the conclusion of the study. The investigators examined four to eight fasted subjects per study morning. Trial visits lasted approximately 45-60 minutes each and took place in the morning (7am-11am). Participants were offered refreshments at the end of their appointment.

If participants wished to be screened for participation in the study, they would receive the Participant Information Sheet and then be checked against the study inclusion and exclusion criteria using a 'Screening Questionnaire' , administered by a member of the D-SOL Research Team by phone or self-reported by email.

Baseline visit:

If eligible, participants were invited for the baseline visit. At this visit, they were first given time to discuss the Participant Information Sheet and any questions they may have regarding the study. Informed consent was discussed and participants were asked to sign the consent form, and offered a copy to keep for themselves.

Baseline procedures:

* Health and Lifestyle questionnaire administered by a member of the D-SOL Research Team.
* Anthropometrics and blood pressure measured, and fasted blood sample taken (serum 25OHD levels, 1,25-dihydroxy vitamin D, serum calcium, albumin, parathyroid hormone, C-terminal telopeptide (CTX) ≈25ml) with an additional ≈10 ml for genetic profiling and ≈15 for storage for future measurements of nutritional markers.
* pQCT scan of the non-dominant forearm (UK trial) or dual energy x-ray absorptiometry (DEXA) scan (Brazil trial).
* Bioelectrical impedance analysis (BIA) for body composition.
* Provision of randomly assigned daily supplement (30 days' supply), food diaries and sunlight dosimeters and sunlight exposure diary to be returned at 12 week visit. Follow-up appointment details arranged.

Final visit

* Final adverse event/compliance interview completed with investigator.
* Daily outdoor exposure diary, food diary and sunlight dosimeter received from participant and checked for consistency at visit.
* Anthropometrics and blood pressure measured, and blood sample taken (serum 25OHD levels, 1,25-dihydroxy vitamin D, serum calcium, albumin, parathyroid hormone, C-terminal telopeptide (CTX) ≈25ml) with an additional ≈10 ml for genetic profiling and ≈15 for storage for future measurements of nutritional markers.
* Bioelectrical impedance analysis (BIA) for body composition.

DNA profiling procedure - After 12 weeks: Selection of participant samples encompassing the best and worst supplementation-responders in each group, subject to previous consent form singed by participant. Vitamin D related genes will be genotyped in DNA isolated from the study blood samples, DNA will be extracted and vitamin D polymorphisms will be determined by University of Surrey's genetic labs.

A trained phlebotomist took the blood samples required as part of the trial protocol. Medical cover was available at all times.

Throughout the duration of the trial, the participants were contacted via telephone on a fortnightly basis to discuss any issues with any adverse event and compliance and to maintain good communication with the participants. In the case of a serious adverse event (SAE) this would be recorded and reported it to both the Sponsor (University of Surrey) and the Surrey Ethics Committee.

The final interview was completed at the final study visit. Participants have also been asked to return any supplements that were missed to confirm compliance.

For University of Surrey participants: A peripheral quantitative computed tomography (pQCT) scan was performed on the participant's non-dominant forearm at the baseline visit, to measure volumetric bone mineral density at the 4% and 66% radial site. This will allow for separate measurements of trabecular volumetric bone mineral density (vBMD) and trabecular area (4% site) and cortical vBMD and cortical area (66% site), as well as strength strain index, a measure of bone strength. pQCT also measures bone geometry alongside bone density. Therefore the muscle cross sectional area can be determined, which is a measure of muscle force, to which bone strength is adapted to. One scan was performed at baseline only and effective exposure doses were between ~1.5-1.8uSv.

For Federal University of Goiás participants: Body composition (absolute and relative amount of lean and fat mass), whole body mineral density and lower spine and femur bone mineral density was measured with the use of DEXA (located at the Nutrition Clinic based at the Federal University of Goiás), at baseline only. Two scans were performed at baseline for each participant: one to assess the whole body mineral density and body composition, and the other to specifically assess fracture risk by scanning the spine and femoral head. Effective exposure doses for theses scans are ~8uSv and ~4uSv respectively.

Results of the body composition, vitamin D status and dietary intake from the self-reported food diaries will be made available to the subjects upon request. The results from the blood analysis will be reported to the subject if there are any health concerns raised. If the results are within healthy ranges the participants will not be contacted unless they specifically request for this information. The investigators will not be contacting their general practitioner (GP) if there are any concerns raised in the study however the investigators will stress that they should contact their GP themselves to discuss the results.

The trial was conducted in compliance with the principles of the Declaration of Helsinki (2008), the principles of Good Clinical Practice and in accordance with The Medicines for Human Use (Clinical Trials) Regulations 2004 and Amended Regulations 2006.

Detailed protocol and supporting documents were submitted for review by the University of Surrey Ethics Committee and the Federal University of Goiás, Brazil. The study received favourable ethical opinion from both Committees prior to commencing the study. Annual progress reports and a final report will be submitted to the ethics committees as defined in their respective regulations.

ELIGIBILITY:
Inclusion Criteria:

Brazilian nationality Living in the UK or in Brazil for more than 2 months

Exclusion Criteria:

* Currently receiving treatment for medical conditions that are likely to affect vitamin D metabolism ( osteoporosis therapy, anti-estrogens treatment, antiepileptic drugs, breast-cancer treatment)
* Hypercalcaemia (>2.5mmol/L) - assessed and excluded at baseline
* Regular use of sun-beds
* Having a holiday trip for more than 4 weeks, one month prior to commencing the study or plans for a holiday trip out of the country of residence within the study period.
* Use of vitamin supplements containing vitamin D (if the prospective participants agrees to stop Vitamin D supplementation to join the study, a wash-out period of 8 weeks prior to commencing the trial would be acceptable).
* Pregnant or planning a pregnancy during the study period.

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline vitamin D status at 12 weeks of vitamin D supplementation | baseline and 12 weeks
  These will be assessed by measuring serum 25(OH)D (in nmol/L) levels in participants at baseline and 12 weeks

SECONDARY OUTCOMES:
Analyze the difference regarding time and intensity of sun exposure between Brazilian women living in Brazil and Brazilian women living in the UK. | baseline
  These will be assessed by participants use of individual sunlight dosimeters and self-reported sun exposure diary
Prevalence of inadequate dietary Vitamin D intake in these women | baseline
  These will be assessed by self-reported food diaries
Baseline prevalence of insufficient/deficient levels of vitamin D in these women. | baseline
  These will be assessed by measuring serum 25(OH)D (in nmol/L) levels in participants at baseline
Change in the number of participants with insufficient/deficient levels of vitamin D after intervention | baseline and after 12 weeks intervention
  These will be assessed by measuring serum 25(OH)D (in nmol/L) levels in participants during winter (baseline and final visit)
Influence of latitude on vitamin D optimal levels. | baseline
  These will be assessed by comparing measurements of serum 25(OH)D (in nmol/L) levels in participants at baseline between women living in the UK (latitude 51 North) and those living in Brazil (latitude 16 South)
Influence of skin pigmentation on vitamin D optimal levels. | baseline
  These will be assessed by comparing baseline measurements of serum 25(OH)D (in nmol/L) levels and self-reported skin type
Vitamin D status influence on bone health | baseline
  Elucidation of the association between Vitamin D status and markers of calcium of calcium metabolism
Vitamin D supplementation response dependence on initial vitamin D levels. | baseline and after 12 weeks intervention
  Assessed by comparing baseline and after intervention measurements of serum 25(OH)D (in nmol/L) levels.
Genetic and enzymatic mechanisms underlying the response to vitamin D supplementation | baseline and after 12 weeks intervention
  These will be assessed by genotyping for polymorphisms related to vitamin D metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Kath Hart, Ph.D, Study Chair — Lecturer, Department of Nutritional Sciences, University of Surrey; Patricia Borges Botelho, Ph.D, Study Chair — Lecturer, Post-graduate Department of Nutrition, Federal University of Goiás; Laura Tripkovic, Ph.D, Study Chair — Teaching Fellow, Department of Nutritional Sciences, University of Surrey
Locations (2):
- Federal University of Goiás, Goiânia, Goiás, Brazil
- University of Surrey, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adams JS, Hewison M. Update in vitamin D. J Clin Endocrinol Metab. 2010 Feb;95(2):471-8. doi: 10.1210/jc.2009-1773. PMID 20133466
- [Background] Bandeira F, Griz L, Freese E, Lima DC, The AC, Diniz ET, Marques TF, Lucena CS. Vitamin D deficiency and its relationship with bone mineral density among postmenopausal women living in the tropics. Arq Bras Endocrinol Metabol. 2010 Mar;54(2):227-32. doi: 10.1590/s0004-27302010000200020. PMID 20485913
- [Background] Lips P. Vitamin D deficiency and secondary hyperparathyroidism in the elderly: consequences for bone loss and fractures and therapeutic implications. Endocr Rev. 2001 Aug;22(4):477-501. doi: 10.1210/edrv.22.4.0437. PMID 11493580
- [Background] Wang TJ, Zhang F, Richards JB, Kestenbaum B, van Meurs JB, Berry D, Kiel DP, Streeten EA, Ohlsson C, Koller DL, Peltonen L, Cooper JD, O'Reilly PF, Houston DK, Glazer NL, Vandenput L, Peacock M, Shi J, Rivadeneira F, McCarthy MI, Anneli P, de Boer IH, Mangino M, Kato B, Smyth DJ, Booth SL, Jacques PF, Burke GL, Goodarzi M, Cheung CL, Wolf M, Rice K, Goltzman D, Hidiroglou N, Ladouceur M, Wareham NJ, Hocking LJ, Hart D, Arden NK, Cooper C, Malik S, Fraser WD, Hartikainen AL, Zhai G, Macdonald HM, Forouhi NG, Loos RJ, Reid DM, Hakim A, Dennison E, Liu Y, Power C, Stevens HE, Jaana L, Vasan RS, Soranzo N, Bojunga J, Psaty BM, Lorentzon M, Foroud T, Harris TB, Hofman A, Jansson JO, Cauley JA, Uitterlinden AG, Gibson Q, Jarvelin MR, Karasik D, Siscovick DS, Econs MJ, Kritchevsky SB, Florez JC, Todd JA, Dupuis J, Hypponen E, Spector TD. Common genetic determinants of vitamin D insufficiency: a genome-wide association study. Lancet. 2010 Jul 17;376(9736):180-8. doi: 10.1016/S0140-6736(10)60588-0. Epub 2010 Jun 10. PMID 20541252
- [Derived] Mendes MM, Hart KH, Williams EL, Mendis J, Lanham-New SA, Botelho PB. Vitamin D Supplementation and Sunlight Exposure on Serum Vitamin D Concentrations in 2 Parallel, Double-Blind, Randomized, Placebo-Controlled Trials. J Nutr. 2021 Oct 1;151(10):3137-3150. doi: 10.1093/jn/nxab209. PMID 34255034

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT03318029/Prot_SAP_000.pdf